CLINICAL TRIAL: NCT04262479
Title: A Pilot Study on Safety, Feasibility and Insulin-promotion by Intra-inguinal Lymph Node Injections of Glutamic Acid Decarboxylase (GAD) in Patients With LADA Type of Diabetes
Brief Title: Injections of Glutamic Acid Decarboxylase (GAD) for LADA Type of Diabetes
Acronym: GADinLADA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Diamyd Medical AB (Industry); Karolinska Institutet (Other); Linkoeping University (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GADinLADA; 2019-002692-34 (EudraCT Number)
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Latent Autoimmune Diabetes in Adults
Keywords: Glutamic Acid Decarboxylase; Alum Compounds; Injections; Inguinal Canal; Diamyd; rhGAD65; Vitamin D
MeSH Terms: conditions — Latent Autoimmune Diabetes in Adults | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GAD-vaccination with vitamin D suppletion (Experimental): Each study participant will receive 3 injections of 4 µg GAD-alum (Diamyd). The first, second and third injection will be one month apart.
  Vitamin D (Divisun 2000 IE) will be given from one month before the first injection of GAD-alum until one month after the third injection (120 days in total).
  Interventions: Drug: recombinant human glutamic acid dehydrogenase (rhGAD65), formulated in aluminium hydrogel; Drug: Vitamin D

INTERVENTIONS:
Drug: recombinant human glutamic acid dehydrogenase (rhGAD65), formulated in aluminium hydrogel — 3 intra-inguinal injections (into the lymph nodes) of GAD-alum one month apart. Supplier Diamyd Medical AB in Stockholm, Sweden
  Other Names: GAD-alum (Diamyd(R))
Drug: Vitamin D — 1 tablet/day, total daily dose of 2000 IE given per os from day -30 through day 90. Supplier Meda, Solna, Sweden
  Other Names: Divisun 2000 IE

SUMMARY:
This study will evaluate the effects of 3 intra-nodal injections of GAD-alum (Diamyd), together with oral vitamin D supplementation. Safety and feasibility of the treatment will be evaluated and also effects on the immune system and on the preservation of endogenous insulin production.

DETAILED DESCRIPTION:
The purpose of the trial is to evaluate the effects of 3 intra-nodal injections of GAD-alum, together with oral vitamin D supplementation, in a population of LADA patients with high GADA titers. Effects will be summarized at 5 and 12 months after the first injection.

* The primary objective is to evaluate safety and feasibility of this treatment regimen.
* Secondary objectives are to test if the treatment induces a strong GAD-specific immune response similar to what has previously been observed in type 1 diabetes patients and to test for indications of preservation of endogenous insulin production.

The study is an open label Phase IIa feasibility trial. It is a pilot study that does not include a placebo arm.

Antidiabetic medication in the form of metformin is acceptable before and during the trial. Study participants must be insulin independent at baseline, but if the need for insulin treatment develops during the trial, such treatment will be given.

GAD-alum will be injected directly into an inguinal lymph node by a qualified radiologist.

Patients will be followed for a total of 12 months during which their endogenous insulin production and immune response will be evaluated at regular intervals throughout the study period. Urine and blood samples will be taken for safety, diabetes status assessments, vitamin D levels and immunological assessments. Concomitant medication and demographics will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by the patient.
2. Diagnosis of LADA and diabetes debut within the last 18 months before inclusion. LADA should be defined by the criteria of age ≥30 years at the onset of diabetes, anti-GAD positivity and no clinical need for permanent insulin treatment during the first 3 months after the diagnosis of diabetes.
3. Fasting C-peptid levels ≥ 0.3 nmol/l
4. High GADA titers (>190 U/ml)
5. Patients must be insulin independent at baseline by clinical judgement and C-peptide criteria
6. Antidiabetic medication in the form of metformin is acceptable for inclusion as well as medications not mentioned under exclusion criteria
7. Females must agree to avoid pregnancy, and must have a negative urine pregnancy test.

Patients of childbearing potential must agree to use adequate contraception, until one (1) year after the last administration of GAD-alum. Adequate contraception is as follows:

For females of childbearing potential:

1. oral (except low-dose gestagen (lynestrenol and norestisteron)), injectable, or implanted hormonal contraceptives
2. combined (estrogen and progestogen containing)
3. oral, intravaginal or transdermal progesterone hormonal contraception associated with inhibition of ovulation
4. intrauterine device
5. intrauterine hormone-releasing system (for example, progestin-releasing coil)
6. bilateral tubal occlusion
7. vasectomized male (with appropriate post vasectomy documentation of the absence of sperm in the ejaculate)
8. male partner using condom
9. abstinence from heterosexual intercourse

For males of childbearing potential:

1. condom (male)
2. abstinence from heterosexual intercourse

Exclusion Criteria:

1. Current or previous treatment with immunosuppressant therapy (topical or inhaled steroids are accepted)
2. Continuous treatment with anti-inflammatory drug (sporadic treatment e.g. because of headache or in connection with fever a few days will be accepted)
3. Systemic treatment with glucocorticoids
4. Treatment with any vaccine, including influenza vaccine, within 1 month prior to planned first study drug dose or planned treatment with any vaccine up to 1 month after the last injection with study drug
5. Antidiabetic medication (metformin excepted)
6. Significantly abnormal hematology results at screening (i.e. anemia with hemoglobin < 12 g/L).
7. A history of epilepsy, head trauma or cerebrovascular accident, or clinical features of continuous motor unit activity in proximal muscles
8. Clinically significant history of acute reaction to vaccines in the past.
9. Renal disease (as defined by serum creatinine >150 µmol/l)
10. Serious cardiovascular events (myocardial infarction, stroke) within the last year preceding recruitment.
11. Participation in other clinical trials with a new chemical entity within the previous 3 months
12. A history of alcohol or drug abuse
13. Known HIV or hepatitis
14. Presence of associated serious disease or condition, including active skin infections that preclude intralymphatic injection, which in the opinion of the investigator makes the patient non-eligible for the study
15. Other serious chronic disease as judged by investigator.
16. Females who are lactating, are pregnant or intend to become pregnant.
17. Inability or unwillingness to comply with the provisions of this protocol
18. Deemed by the investigator not being able to follow instructions and/or follow the study protocol
19. Treatment any other supplementation of with vitamin D, marketed or not, or unwilling to abstain from such medication during the trial 120 days daily intake of Divisun (non-investigational medicinal product)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Hildur Henriksen, MD PhD, Study Director — St Olavs Hospital, Medisinsk Klinikk; Torstein Baade Rø, MD, Study Director — Norwegian University of Science and Technology, IKOM
Locations (2):
- Department of Endocrinology, St Olavs Hospital, Trondheim, Norway
- Akademiskt Specialistcentrum, Centrum for Diabetes, and Karolinska Institute, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Hals IK, Fiskvik Fleiner H, Reimers N, Astor MC, Filipsson K, Ma Z, Grill V, Bjorklund A. Investigating optimal beta-cell-preserving treatment in latent autoimmune diabetes in adults: Results from a 21-month randomized trial. Diabetes Obes Metab. 2019 Oct;21(10):2219-2227. doi: 10.1111/dom.13797. Epub 2019 Jun 19. PMID 31148332

RESULTS

PARTICIPANT FLOW:
Groups:
- GAD-vaccination With Vitamin D Suppletion: Each study participant will receive 3 injections of 4 µg GAD-alum (Diamyd). The first, second and third injection will be one month apart.
  Vitamin D (Divisun 2000 IE) will be given from one month before the first injection of GAD-alum until one month after the third injection (120 days in total).
  recombinant human glutamic acid dehydrogenase (rhGAD65), formulated in aluminium hydrogel: 3 intra-inguinal injections (into the lymph nodes) of GAD-alum one month apart.
  Supplier Diamyd Medical AB in Stockholm, Sweden
  Vitamin D: 1 tablet/day, total daily dose of 2000 IE given per os from day -30 through day 90. Supplier Meda, Solna, Sweden
Period: Overall Study
Arm/Group | GAD-vaccination With Vitamin D Suppletion
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GAD-vaccination With Vitamin D Suppletion
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 46 [30 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 8
  Norway | 6
Time from diagnosis to inclusion, months [Median (Full Range); unit: months] | 4 [3 to 15]
BMI, kg/m^2 [Median (Full Range); unit: kg/m^2] | 25.1 [19.2 to 36.7]
Fasting C-peptide, nmol/L [Median (Full Range); unit: nmol/L] | 0.55 [0.25 to 1.35]
Fasting glucose, mmol/L [Median (Full Range); unit: mmol/L] | 6.7 [4.8 to 12.5]
HbA1c, mmol/mol [Median (Full Range); unit: mmol/mol] | 42 [35 to 65]

OUTCOME MEASURES:

1. Primary Outcome: Injection Site Skin Reactions
Description: Injection site skin reactions 1 hour post injection, i.e., erythema, oedema, haematoa, tenderness, pain, itching or other finding.
Time Frame: 1 hour
Population: All study participants received 3 injections of 4 µg GAD-alum.
Measure: Number; unit: events
Arm/Group | GAD-vaccination With Vitamin D Suppletion
Number analyzed (Participants) | 14
events | 4

2. Primary Outcome: Occurrence of Adverse Events (AEs) During 5 Months From Baseline.
Description: AEs were continuously monitored and registered from the baseline visit (first injection of GAD-alum) to the end of study (12 months after the baseline visit). The total number of AEs registered for all 14 participants during the first 5 months from baseline was summarized when all 14 participants had completed their 5 months study visit (i.e., 5 months after the baseline visit). At the end of study, when all 14 participants had completed their 12 months study visit, the total number of AEs registered for all 14 participants during the 12 months from baseline was summarized.
Time Frame: From baseline (first injection of GAD-alum) to 5 months after baseline.
Measure: Number; unit: AEs
Arm/Group | GAD-vaccination With Vitamin D Suppletion
Number analyzed (Participants) | 14
AEs | 28
Statistical Analysis 1: Comparison: GAD-vaccination With Vitamin D Suppletion; Test type: Other; Counting number of events

3. Primary Outcome: Occurrence of Adverse Events (AEs) During the Study.
Description: AEs were continuously monitored and registered from the baseline visit (first injection of GAD-alum) to the end of study (12 months after the baseline visit/first injection of GAD-alum). The total number of AEs registered for all 14 participants during the first 5 months from baseline was summarized when all 14 participants had completed their 5 months study visit (i.e., 5 months after the baseline visit). At the end of study, when all 14 participants had completed their 12 months study visit, the total number of AEs registered for all 14 participants during the 12 months from baseline was summarized.
Time Frame: From baseline (first injection of GAD-alum) to 12 months after baseline.
Measure: Number; unit: AEs
Arm/Group | GAD-vaccination With Vitamin D Suppletion
Number analyzed (Participants) | 14
AEs | 34
Statistical Analysis 1: Comparison: GAD-vaccination With Vitamin D Suppletion; Test type: Other; Counting number of events

4. Primary Outcome: Serum GAD65A Titers, Change From Baseline at 5 Months After Baseline.
Description: Values present changes in serum GAD65A titers from baseline (first injection of GAD-alum) to 5 months after baseline.
  Calculation: Value at 5 months minus value at baseline.
Time Frame: Baseline (first injection of GAD-alum) and 5 months after baseline.
Measure: Median (Full Range); unit: U/mL
Arm/Group | GAD-vaccination With Vitamin D Suppletion
Number analyzed (Participants) | 14
U/mL | 59218 [-2800 to 1006000]
Statistical Analysis 1: Comparison: GAD-vaccination With Vitamin D Suppletion; Test type: Other; p < 0.001, Wilcoxon signed rank test — P-value threshold for significance: <0.05

5. Primary Outcome: Serum GAD65A Titers, Change From Baseline at 12 Months After Baseline.
Description: Values present changes in serum GAD65A titers from baseline (first injection of GAD-alum) to 12 months after baseline.
  Calculation: Value at 12 months minus value at baseline.
Time Frame: Baseline and 12 months after baseline.
Measure: Median (Full Range); unit: U/mL
Arm/Group | GAD-vaccination With Vitamin D Suppletion
Number analyzed (Participants) | 14
U/mL | 26082 [-631000 to 87455]
Statistical Analysis 1: Comparison: GAD-vaccination With Vitamin D Suppletion; Test type: Other; p < 0.05, Wilcoxon signed rank test — P-value threshold for significance: <0.05

6. Secondary Outcome: Insulin Secretion, Change From Baseline to 5 Months After Baseline.
Description: Values present changes in serum values of glucagon-stimulated C-peptide from baseline (first injection of GAD-alum) to 5 months after baseline.
  Calculation: Value at 5 months minus value at baseline.
Time Frame: Baseline (first injection of GAD-alum) and 5 months after baseline.
Measure: Median (Full Range); unit: nmol/L
Arm/Group | GAD-vaccination With Vitamin D Suppletion
Number analyzed (Participants) | 14
nmol/L | 0.00 [-0.50 to 0.70]
Statistical Analysis 1: Comparison: GAD-vaccination With Vitamin D Suppletion; Test type: Other; p < 0.61, Wilcoxon signed rank test — P-value threshold for significance: <0.05

7. Secondary Outcome: Insulin Secretion, Change From Baseline to 12 Months After Baseline.
Description: Values present changes in serum values of glucagon-stimulated C-peptide from baseline (first injection of GAD-alum) to 12 months after baseline.
  Calculation: Value at 12 months minus value at baseline.
Time Frame: Baseline (first injection of GAD-alum) and 12 months after baseline.
Measure: Median (Full Range); unit: nmol/L
Arm/Group | GAD-vaccination With Vitamin D Suppletion
Number analyzed (Participants) | 14
nmol/L | -0.10 [-0.60 to 0.70]
Statistical Analysis 1: Comparison: GAD-vaccination With Vitamin D Suppletion; Test type: Other; p < 0.30, Wilcoxon signed rank test — P-value threshold for significance: <0.05

8. Secondary Outcome: Change in HbA1c
Description: HbA1c at 12 months vs. baseline (first injection)
Time Frame: from baseline to 12 months after the first injection
Measure: Median (Full Range); unit: mmol/mol
Arm/Group | GAD-vaccination With Vitamin D Suppletion
Number analyzed (Participants) | 14
mmol/mol | 3.0 [-1.0 to 28.0]
Statistical Analysis 1: Comparison: GAD-vaccination With Vitamin D Suppletion; Test type: Other; p < 0.002, Wilcoxon signed rank test — P-value threshold for significance: <0.05

9. Secondary Outcome: Change in Fasting Glucose
Description: Change in fasting glucose at 12 months vs baseline (first injection)
Time Frame: From baseline to 12 months after the first injection
Measure: Median (Full Range); unit: mmol/L
Arm/Group | GAD-vaccination With Vitamin D Suppletion
Number analyzed (Participants) | 14
mmol/L | -0.05 [-1.00 to 3.10]
Statistical Analysis 1: Comparison: GAD-vaccination With Vitamin D Suppletion; Test type: Other; p < 0.72, Wilcoxon signed rank test — P-value threshold for significance: <0.05

10. Secondary Outcome: Change in Fasting C-peptide
Description: Change in fasting glucose at 12 months vs baseline (first injection)
Time Frame: Between baseline and 12 months after the first injection
Measure: Median (Full Range); unit: nmol/L
Arm/Group | GAD-vaccination With Vitamin D Suppletion
Number analyzed (Participants) | 14
nmol/L | -0.03 [-0.25 to 0.05]
Statistical Analysis 1: Comparison: GAD-vaccination With Vitamin D Suppletion; Test type: Other; p < 0.03, Wilcoxon signed rank test — P-value threshold for significance: <0.05

11. Secondary Outcome: Change in Maximum C-peptide During Mixed Meal Tolerance Test (MMTT)
Description: Change in maximum C-peptide value at 12 months vs baseline (first injection)
Time Frame: between baseline 12 months after the first injection
Measure: Median (Full Range); unit: nmol/L
Arm/Group | GAD-vaccination With Vitamin D Suppletion
Number analyzed (Participants) | 14
nmol/L | -0.30 [-0.90 to 0.50]
Statistical Analysis 1: Comparison: GAD-vaccination With Vitamin D Suppletion; Test type: Other; p < 0.044, Wilcoxon signed rank test — P-value threshold for significance: <0.05

12. Primary Outcome: Serum GAD65A Titers, Change From Baseline at 12 Months After Baseline.
Description: as for outcome 5
Time Frame: Baseline (first injection of GAD-alum) and 12 months after baseline.
Measure: Median (Full Range); unit: U/mL
Arm/Group | GAD-vaccination With Vitamin D Suppletion
Number analyzed (Participants) | 14
U/mL | 26082 [-631000 to 87455]

ADVERSE EVENTS:
Time Frame: One year. AEs were continuously monitored and registered from the baseline visit (first injection of GAD-alum) to the end of study (12 months after the baseline visit/first injection of GAD-alum).
Arm/Group | GAD-vaccination With Vitamin D Suppletion
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GAD-vaccination With Vitamin D Suppletion (N=14)
Angina unstable (Cardiac disorders) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GAD-vaccination With Vitamin D Suppletion (N=14)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Vertigo or vertigo positional (Ear and labyrinth disorders) | 2 (2)
diarrhoea (Gastrointestinal disorders) | 2 (2)
Pancreatic cystadenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
General disorders and administration site conditions (General disorders) | 6 (8) — Chest pain, injection site erythema or haemorrhage or pain, pyrexia,
Biliary colic (Hepatobiliary disorders) | 1 (1)
COVID-19, nasopharyngitis, upper respiratory tract infection (Infections and infestations) | 6 (6)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1)
Wrong product administered (Injury, poisoning and procedural complications) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Blood urine present (Investigations) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (3)
Nasal congestion and throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Menopause (Social circumstances) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/79/NCT04262479/Prot_SAP_000.pdf